CLINICAL TRIAL: NCT04763941
Title: Reliability of the Clinical Dementia Rating Scale From the Medical Record in Comparison With the Reference Method.
Brief Title: Clinical Dementia Rating Medical Record
Acronym: CLIMER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0508
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-01

CONDITIONS: Clinical Dementia Rating (CDR) From the Analysis of Medical Record; Clinical Dementia Rating (CDR) Face-to-face Interview With the Patient
Keywords: CDR; memory consultation; patient's file; reliability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Memory consultation patient: The study will be conducted on the basis of the patient consulting in Memory Consultation, specifically with the information already collected in normal care and the MEMORA cohort.
  Interventions: Diagnostic Test: CDR assessment face-to-face

INTERVENTIONS:
Diagnostic Test: CDR assessment face-to-face — The assessment of the CDR is administered once by a psychologist with the patient and his caregiver.

SUMMARY:
The assessment of severity of the cognitive and functional impairment is essential in the follow-up of patients with neurocognitive disorders and in the assessment of the effectiveness of therapeutics. However, the systematic assessment of the Clinical Dementia Rating (CDR) scale is limited due to the time required to complete it (approximately 45 min to 1 hour). Insofar as studies have shown correspondences between the CDR and scales measuring cognitive and neuropsychological performance, and as part of memory consultations, several functional and neuropsychological scales are systematically administered, we wish to conduct a study validating the feasibility of the CDR based on information already available in the patient's file compared to the evaluation of the CDR by the usual method (face-to-face interview in consultation).

This study should highlight the feasibility of scoring the CDR-SB from the files of patients in memory consultation, first in terms of reliability of the scores obtained compared to the standard evaluation, and on the other hand in terms of organization and duration of administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has CDR assessment in face-to-face interview during the memory consultation,
* Patient with an isolated cognitive complaint or a neurocognitive disorder
* Patient included in the MEMORA cohort

Exclusion Criteria:

* Patient or caregiver who does not wish their data to be used for research purposes within the framework of the MEMORA cohort.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will be conducted on the basis of the patient consulting in Memory Consultation, specifically with the information already collected in normal care and the MEMORA cohort.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
CDR Sum of boxes (CDR-SB) score out of 18 | The CDR-SB score is collected at the baseline.
  The CDR-SB score is obtained in normal condition and on file for the same patients. The CDR-SB score makes it possible to distinguish the following classes: 0 (normal), 0.5-4 (questionable cognitive impairment), 0.5-2.5 (questionable impairment), 3-4 (very mild major TNC or very mild dementia), 4.5- 9 (mild or mild dementia), 9.5-15.5 (moderate dementia), 16-18 (severe dementia).
  The patient's aptitudes are assessed in 6 different areas: 3 cognitive skills: memory, orientation and judgment, 3 acts of everyday living: participation in collective life, home occupations and hobbies, personal care.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bathsavanis, Psy D, Study Director — Hôpital des Charpennes; Pierre Krolak-Salmon, MD, Principal Investigator — Hopital Edouard Herriot
Locations (1):
- Hôpital Des Charpennes, Villeurbanne, France

REFERENCES:
- [Derived] Dauphinot V, Calvi S, Moutet C, Xie J, Dautricourt S, Batsavanis A, Krolak-Salmon P, Garnier-Crussard A. Reliability of the assessment of the clinical dementia rating scale from the analysis of medical records in comparison with the reference method. Alzheimers Res Ther. 2024 Sep 5;16(1):198. doi: 10.1186/s13195-024-01567-9. PMID 39238042